CLINICAL TRIAL: NCT06405256
Title: Displacement and Deformation Analysis of Adaptive Radiotherapy Based on MR-Linac for Large Brain Metastases
Brief Title: Magnetic Resonance Imaging-guided Adaptive Radiotherapy for Large Brain Metastases
Status: Recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: BMMRIgART
Record Dates: First submitted 2024-05-04; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-03

CONDITIONS: Brain Metastases
Keywords: Magnetic Resonance Imaging-guided Adaptive Radiotherapy
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BM patients receiving MRIgART: For it's an observational study, all patients eligible will be divided into the group "BM patients receiving MRIgART"
  Interventions: Radiation: magnetic resonance imaging-guided adaptive radiotherapy

INTERVENTIONS:
Radiation: magnetic resonance imaging-guided adaptive radiotherapy — Stereotactic Radiotherapy (with the prescribed dose of PTV 52-52.5 Gy, 13-15 fractions and Boost (if any) 60Gy, 15 fractions)

SUMMARY:
This study is an ambispective cohort study to evaluate the displacement and deformation of large brain metastases (BM) treated with magnetic resonance imaging-guided adaptive radiotherapy (MRIgART)

DETAILED DESCRIPTION:
All patients had a pathologically confirmed malignant cancer and were diagnosed with brain metastases (BM) by enhanced magnetic resonance imaging (MRI) with BM volume of 2cm and above. All patients received Unity MR-linac adaptive radiotherapy. Gross tumor volume (GTV) and organs at risk (OARs) were re-delineated for every image set and analyzed for displacement and deformation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years; KPS score ≥ 60.
2. pathologically confirmed lung cancer.
3. diagnosed with brain metastases by enhanced MRI.
4. BM volume ≥ 2cm.
5. Anticipated time to survival>3 months.
6. Treated with Unity MR-linac.
7. Good compliance; Able to stay still in supine position for 45 minutes and above.

Exclusion Criteria:

1. Fail to complete radiotherapy as planned; Anticipated time to survival less than 3 months.
2. Suffer from severe back pain in supine position, unable to receive Unity MR-linac.
3. Suffer from severe claustrophobia.
4. Incomplete pre-Unity image data.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients from Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-01-03 (Actual); Primary Completion 2025-03-18 (Estimated); Study Completion 2025-03-18 (Estimated)

PRIMARY OUTCOMES:
Intra-cranial progression-free survival (IPFS) | From the date of radiation until the date of first documented intracalcarine recurrence or progression, or date of death from any cause, whichever came first, assessed up to 12 months.
  Defined as the time from date of radiation until the date of first documented intracalcarine recurrence or progression, or date of death from any cause, whichever came first.

SECONDARY OUTCOMES:
Local control rate (LCR) | Tumor assessment using RECIST will be performed at baseline then every 3 months from first treatment until objective progression or death from any cause, assessed up to 12 months.
  LCR will be calculated as the number of patients without intrathoracic tumor progression per RECIST Criteria.
Overall survival (OS) | From the date of radiation until the date of any documented death due to any cause,, assessed up to 12 months.
  Defined as the time from the date of radiation to the date of any documented death due to any cause.
Objective Response Rate (ORR) | Tumor assessment using RECIST will be performed at baseline then every 3 months from first treatment until objective progression or death from any cause, assessed up to 12 months.
  The objective response rate (ORR) will be calculated as the number of patients with CR or PR per RECIST Criteria.
  Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Disease control rate (DCR) | Tumor assessment using RECIST will be performed at baseline then every 3 months from first treatment until objective progression or death from any cause, assessed up to 12 months.
  DCR will be calculated as the number of patients with CR, PR or sustained SD≥6 weeks per RECIST Criteria.
  Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase.
Adverse Event | AEs and SAEs must be collected from the start of treatment to 28 days after discontinuation of radiation, up to 12 months.
  The incidence of adverse events (AEs) and serious adverse events (SAEs) is evaluated by EORTC/RTOG Radiation Grading System Criteria and CTCAE 5.0. Appropriate description of AEs and laboratory data/vital signs will be produced. Number of patients who had at least one adverse event will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Nan Bi, MD, Principal Investigator — Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Chinese Academy of Medical Science and Peking Union Medical College, Beijing, China